CLINICAL TRIAL: NCT04785443
Title: Contribution of Indocyanine Green Angiography in the Detection of Parathyroids and the Prevention of Hypoparathyroidism Post Total Thyroidectomy
Brief Title: Contribution of ICG Angiography in the Detection of Parathyroids and the Prevention of Hypoparathyroidism Post Total Thyroidectomy
Acronym: HYPOCAAVI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 29BRC20.0208
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Thyroid Diseases
Keywords: Hypocalcemia; Hypoparathyroidism; Angiography
MeSH Terms: conditions — Thyroid Diseases; Hypocalcemia; Hypoparathyroidism | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Monocentric, comparative, randomized, single-blind, controlled trial against the reference method
Who Masked: Participant
Masking Description: Simple blind (only participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG group (Experimental): Patient receiving 2 or 3 intraoperative injections of indocyanine green.
  Interventions: Drug: ICG
- Control group (Other): Patient benefiting from the traditional surgical act
  Interventions: Procedure: Control group

INTERVENTIONS:
Drug: ICG — During thyroidectomy surgery, the patient will received 2 or 3 injections of 5 mg as a bolus. The first one during the dissection of the first lobe, then during the dissection of the second lobe and finally if needed, a 3rd injection will be done at the end of the dissection.
  Patients will then be followed during 6 months.
  Arms: ICG group
Procedure: Control group — During thyroidectomy surgery, patients are treated according to traditional surgery with detection of parathyroids with the naked eyes.
  Patients will then be followed during 6 months.
  Arms: Control group

SUMMARY:
* Hypoparathyroidism is the most common complication after a total thyroidectomy surgery. It becomes permanent after 6 months.
* Untreated permanent hypoparathyroidism is a source of numerous complications in general and therefore requires lifelong replacement therapy resulting in a significant deterioration in quality of life.
* The intraoperative use of indocyanine green (ICG) angiography has recently been described as a reliable means of detecting parathyroidism and predicting the risk of postoperative hypoparathyroidism.
* This use could prove to be a way to preserve parathyroid in vivo and thus reduce post-operative hypoparathyroidism rates.

DETAILED DESCRIPTION:
Hypoparathyroidism is the most common complication after a total thyroidectomy surgery. It is most often transient but can sometimes be permanent when it persists for more than 6 months after surgery. The rates are variable, of the order of 32% for transient hypoparathyroidism and 1% for definitive hypoparathyroidism. Untreated permanent hypoparathyroidism is the source of many complications in general and therefore requires lifelong replacement therapy. The result is a significant deterioration in quality of life.

The mechanisms responsible for hypoparathyroidism during thyroidectomy are direct damage to the parathyroid glands, involuntary excision of these glands, and devascularization of these glands.

The detection of parathyroid glands and the prevention of hypoparathyroidism after thyroidectomy therefore represents a major challenge.

The intraoperative use of indocyanine green angiography has recently been described as a reliable means of detecting parathyroid and predicting the risk of postoperative hypoparathyroidism.

In addition, prior studies and intraoperative observations suggest that indocyanine green angiography during thyroid surgery may be a means of preserving parathyroid in vivo and thus reducing post-operative hypoparathyroidism rates.

ELIGIBILITY:
Inclusion Criteria:

* Patient having to undergo a total thyroidectomy
* Signed consent
* Patient beneficiary of a social security regimen

Exclusion Criteria:

* Minor patient under 18 years old
* Major patient protected by law or unable to give informed consent
* Pregnant or breastfeeding woman
* Thyroidectomy totalization
* History of thyroid or parathyroid surgery
* Participation refusal
* Known allergy to ICG
* Woman of child-bearing age not using adequate method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Compare the frequency of albumin-corrected hypocalcemia (blood sugar below 2 mmol/L, a sign associated with hypoparathyroidism) postoperatively between the ICG group and the control group. | Day 2
  Frequency of albumin-corrected hypocalcemia (≤2 mmol/L) within 48 hours postoperatively.

SECONDARY OUTCOMES:
Evaluate the contribution of ICG angiography in the modification of the rate of definitive hypoparathyroidism after total thyroidectomy. | Day 8, Month 1 and Month 6
  Occurrence (yes/no) of albumin-corrected (<2mmol/L) postoperative hypocalcemia at D8, M1 and M6
Determine the contribution of indocyanine green angiography (ICG) during the total thyroidectomy procedure for in vivo detection and preservation of parathyroid glands. | Day 0
  Modification (yes/no) of the surgical procedure by improving the detection of parathyroids or their vascularization during thyroidectomy with the use of indocyanine green angiography.
To evaluate the contribution of indocyanine green angiography in the prediction of postoperative hypocalcemia. | Day 0
  Intraoperative parathyroid vitality score (0=devascularized parathyroid gland to 2 = vascularized thyroid gland) when using indocyanine green angiography.
To determine the interest of indocyanine green angiography (ICG) in the prediction of hypoparathyroidism after total thyroidectomy. | Day 1 and Day 2
  Occurrence (yes/no) of hypo parathormone at D1 and D2 postoperatively (<10ng/L).
Compare the frequency of postoperative hypocalcemia, according to its grade (mild, moderate and deep), between the ICG group and the control group. | D1 and D2
  Frequency of mild (asymptomatic and >1.7mmol/l), moderate (symptomatic and >1.7mmol/l) and profound (<1.7mmol/l) hypocalcemia within 48 hours postoperatively.
Evaluate the tolerance of indocyanine green. | Day 1, Day 2, Day 10
  Occurrence of an adverse event related to the injection of indocyanine green.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe LECLERE, PhD, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion.
Access Criteria: Data access request will be reviewed by the internal committee of Brest University Hospital. Requestor will be required to sign and complete a data access agreement.